CLINICAL TRIAL: NCT05588856
Title: Doctor-patient Partnerships: the Key to a Better Standard of Medical Advice?
Status: Recruiting | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/2354
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Doctor-Patient Relation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Chronic Lung Disease
  Interventions: Other: In depth Interview
- Healthcare professionals
  Interventions: Other: In depth Interview

INTERVENTIONS:
Other: In depth Interview — In depth Interviews

SUMMARY:
Background: The current legal standard of advice in Singapore has three components: distinction of advice from the other parts of clinical consultation (i.e. diagnosis and treatment) for the purpose of standard setting, categories of information that need to be disclosed to patients and how the adequacy of this information is judged in court. A review of empirical data shows that information deficit is not the only or most pressing concern in decision-making from the patients' perspective. The data also reflects the value that is placed on relationships that patients have with their treating doctors. Features of a good doctor-patient relationship can be found in partnerships, which are based on therapeutic alliance and mutuality.

Objective: To develop a contextual understanding of the role of clinical partnerships in Singapore, empirical data is needed from both patients and healthcare workers on their understanding and interpretation of doctor-patient partnerships and how medical decisions are made using this relationship.

Design: A qualitative study using interpretive analysis of semi-structured interviews conducted via in-person, telephone and videoconferencing interviews.

DETAILED DESCRIPTION:
Doctor-patient partnerships: the key to a better standard of medical advice?

Background: The current legal standard of advice in Singapore has three components: distinction of advice from the other parts of clinical consultation (i.e. diagnosis and treatment) for the purpose of standard setting, categories of information that need to be disclosed to patients and how the adequacy of this information is judged in court. A review of empirical data shows that information deficit is not the only or most pressing concern in decision-making from the patients' perspective. The data also reflects the value that is placed on relationships that patients have with their treating doctors. Features of a good doctor-patient relationship can be found in partnerships, which are based on therapeutic alliance and mutuality.

Objective: To develop a contextual understanding of the role of clinical partnerships in Singapore, empirical data is needed from both patients and healthcare workers on their understanding and interpretation of doctor-patient partnerships and how medical decisions are made using this relationship.

Design: A qualitative study using interpretive analysis of semi-structured interviews conducted via in-person, telephone and videoconferencing interviews.

Setting: Singapore General Hospital inpatients and outpatients from Dept of Respiratory and Critical Care Medicine.

Participants:

1. Patients with known chronic lung disease such as Chronic Lung Disease (n=200)
2. Healthcare professionals (eg. doctors and nurses) involved in the management of the above patients (n=100)

   Recruitment:

   Recruitment of all participants will be through the Singapore General Hospital ambulatory clinic or general ward.

   All patients must have a confirmed diagnosis of the chronic lung disease that is consistent with international guidelines. The diagnosis will be verified by the managing physician Informed consent forms will be signed. We will aim for purposive and maximum variation sampling.

   Interview:

   Semi-structured interviews with patients with chronic lung disease and healthcare providers according to the interview guide.

   Each interview will be 45 - 120 minutes during their consultation waiting time, conducted in a counselling/private room is done in person. If participant is agreeable the interviews can be conducted via telephone or videoconferencing.

   All interviews will be audio recorded. The video component of videoconferencing will be deleted.

   The initial interviews will be conducted >1 investigator to ensure standardization of the process.

   We will ask the participants for permission for follow-up interviews and questions.

   We will ask participants to recommend other participants to facilitate snowball sampling especially for the healthcare professionals.

   Data analysis:

   The interview analysis will follow an iterative process (deductively and inductively) All non-English interviews will be translated All interviews will be transcribed before analysis After being transcribed, the audio recordings will be destroyed Coded transcripts will be stored in a password protected computer of the investigators.

   Member checking of transcripts and representative quotes will be allowed.

   Interview Guide (Patients) Examples of questions to guide interview

   Medical condition 1. Describe your medical diagnosis and prognosis 2. Describe your lung condition 3. How will your disease progress? 4. How has this disease impacted your life?

   Decision-making 5. Describe the medical decisions that that you have had to make 6. Share examples of good and less good decision-making experiences 7. Do your healthcare providers support your decision-making? 8. Do you feel that you are in control of your medical decisions? If so why? 9. Are you satisfied with the current medical decision-making process?

   Relationships 10. Describe the relationships that you have had with your healthcare providers 11. Share good (and bad) features of the working relationship with your healthcare providers 12. What should be the aim of the doctor-patient/nurse-patient relationship? 13. What should the healthcare providers goals be for the relationship? 14. What should be your goals for the relationship? 15. Do you feel respected by your healthcare providers? 16. What do you value in your healthcare providers? 17. What makes you satisfied with your doctors? 18. Do your healthcare providers address your concerns?

   Decision-making responsibility 19. Have you got any thoughts about who has responsibility for the decisions that have been made? 20. Who is responsible for the medical decisions that have been made? 21. Who is responsible for the medical decisions when something goes wrong? 22. Who should be making medical decisions for you? 23. Who makes decisions on your behalf?

   Scope of advice 24. What information would you want to make medical decisions? 25. What type of risks would you want to know about before making decisions? 26. Do you want to be told of alternatives before making any medical decision? 27. Who do you think should determine the standard of medical advice? 28. Do you understand the information that you have been given on your medical condition?

   Concerns 29. What are your current concerns and challenges? 30. What does living well mean for you now? 31. What goals do you have when you make medical decisions?

   Informed Consent 32. What do you want to be told before you provide informed consent? 33. Do you find giving informed consent stressful? If so, why? 34. Is informed consent part of the medical encounter or a legal requirement? 35. What is the average you spend speaking to your healthcare provider during each encounter? 36. Would you want to know all the risks about procedures? 37. Would you want to know about very rare but dangerous risks? 38. Would you still want to know the risks even if it may confuse you? 39. How should it be determined if you have been told the right amount of information before making a decisions?

   Goals 40. Do your healthcare providers elicit your beliefs and values? 41. Do those who make decisions on your behalf elicit your beliefs and values? 42. What do you value or want from healthcare? 43. What do you value during your consultation?

   Interview Guide (Healthcare Professionals) Examples of questions to guide interview

   Medical Service 1. Describe how you are involved in the care of patients with this type of chronic lung disease 2. How long have been caring for such patients 3. What training have received in the care of these patients?

   Decision-making 4. Describe the medical decisions that that you have had to make 5. Share examples of good and less good decision-making experiences 6. Do patients expect you to make medical decisions on their behalf? 7. Do you want to make medical decisions on behalf of competent patients? Why? 8. Do you feel that patients are in control of their medical decisions? If so why? 9. Are you satisfied with the current medical decision-making process?

   Relationships 10. Describe the relationships that you have had with your patients 11. Share good (and bad) features of the working relationship with your patients 12. What should be the aim of the doctor-patient/nurse-patient relationship? 13. What should the healthcare providers' goals be for the relationship? 14. What should the patients' goals be for the relationship? 15. Do you feel respected by your patients? 16. What do you value in your relationships with patients?

   Decision-making responsibility 17. Have you got any thoughts about who has responsibility for the decisions that have been made? 18. Who is responsible for the medical decisions that have been made? 19. Who is responsible for the medical decisions when something goes wrong? 20. What is your understanding of the legal position of decision-making responsibility? 21. What is your understanding of the ethical position of decision-making responsibility?

   Scope of advice 22. What information should you give to help patients make medical decisions? 23. What type of risks do you think patients would want to know about before making decisions? 24. Do you want patients want to be told of alternatives before making any medical decision? 25. Who do you think should determine the standard of medical advice? 26. Do you think patients understand the information that they have been given on their medical condition?

   Concerns 27. What are your current concerns and challenges about medical decision-making and professional relationship with patients? 28. What do you think living well mean for your patient? 29. What goals do you have when you make medical recommendations?

   Informed Consent 30. What do you think patients should to be told before they provide informed consent? 31. Do you find taking informed consent stressful? If so, why? 32. Is informed consent part of the medical encounter or a legal requirement? 33. What is the average time you spend speaking to your patient during each encounter? 34. Would your patient want to know all the risks about procedures? 35. Would your patient want to know about very rare but dangerous risks? 36. Would your patient still want to know the risks even if it may confuse them? 37. How should it be determined if your patient has been told the right amount of information before making a decisions?

   Goals 38. Do your elicit your patients beliefs and values before making recommendations? 39. Are the goals of the patient consistent with the goals of medicine? 40. What do your patients value or want from healthcare? 41. What do your patients value or want from the consultation?

   Data extraction

   Data from electronic medical records for patients who have consented to the interview:
   * Age, education, race, religion, occupation
   * Risk factors: Smoking status
   * Co-morbidities: Depression score (PHQ-9) (if applicable)
   * Clinical Scores: eg. BODE, CAT, ACT (if applicable)
   * Medical history, duration and objective severity of lung disease: whether the patient is on long term oxygen, been admitted to ICU and number of exacerbations per year.
   * Any previous ACP counselling: Yes or No or Unsure

   Data from Healthcare workers
   * Age, education, race, religion
   * Designation, profession, years of service in SingHealth, years of service in the profession
   * Formal training in communication and ethics

ELIGIBILITY:
Inclusion Criteria:

* Recruitment of all participants will be through the Singapore General Hospital ambulatory clinic or general ward.

All patients must have a confirmed diagnosis of the chronic lung disease that is consistent with international guidelines. The diagnosis will be verified by the managing physician Informed consent forms will be signed. We will aim for purposive and maximum variation sampling.

Exclusion Criteria:

* None of the above

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic lung disease and healthcare professionals who care for them
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Descriptions of decision-making and relationships | 5 years
  As above

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plans to share data